CLINICAL TRIAL: NCT04084028
Title: Examining Cooking as a Health Behavior in College Students
Brief Title: Cooking as a Health Behavior in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Lizzy Pope, Assistant Professor and DPD Director, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS #00000397; VT-H02510 (Other Grant/Funding Number: USDA Hatch Act Funds)
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Diet, Healthy
Keywords: food agency; cooking
MeSH Terms: interventions — Cookbooks as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Cooking +meal kits and recipes (Experimental): Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal.
  Following 6 weeks of cooking classes, participants will receive 6 weeks of home-delivered meal kits. Following 6 weeks of meal kits, participants will received 6 weeks of recipes. Both the meal kits and recipes will accommodate major dietary needs (vegan, gluten-free, etc.)
  Interventions: Behavioral: Active Cooking Classes; Behavioral: Meal Kits; Behavioral: Recipes
- Active cooking only (Active Comparator): Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal. Unlike the previous arm, no further instruction will be given once cooking classes end.
  Interventions: Behavioral: Active Cooking Classes
- Meal Kits only (Active Comparator): Participants will receive weekly meal kit deliveries for 6 weeks. Following 6 weeks of meal kit deliveries, students will receive emails at the beginning of each week providing them with 5 healthy recipes.
  Interventions: Behavioral: Meal Kits; Behavioral: Recipes
- Control (No Intervention): Participants will receive no interventions.

INTERVENTIONS:
Behavioral: Active Cooking Classes — 6 cooking classes will be held every week for 6 consecutive weeks. The lessons are patterned after Dr. Amy Trubek's cooking pedagogy and will be tailored for those cooking for themselves for the first time. Classes begin with a brief lecture on the day's topic. Students will work in teams of 2 in the foods lab to actively practice skills and cook a meal. Students receive recipes and information sheets that cover pantry supplies, grocery lists, knife skills and cooking equipment. All students attend a 2 hour kitchen intensive demonstration as an orientation.
  Arms: Active Cooking +meal kits and recipes; Active cooking only
Behavioral: Meal Kits — Students receive 6 weeks of home delivered meal kits. Meal kits include ingredients and detailed instructions for 3 meals, which each serve two people. Students may select meals from a list of 18 options that include vegan, vegetarian, and gluten free options.
  Arms: Active Cooking +meal kits and recipes; Meal Kits only
Behavioral: Recipes — Students are emailed a set of recipes once a week for 6 weeks. Recipes include options for breakfast, lunch, dinner, and snacks. Recipe sets include vegan, vegetarian, and gluten-free options. This intervention was cancelled by COVID-related disruptions and did not take place.
  Arms: Active Cooking +meal kits and recipes; Meal Kits only

SUMMARY:
Students who live off campus at the University of Vermont will be recruited to participate in the study which will begin in Fall 2019 and run through May 2020. The intervention is a randomized-controlled trial where students will be randomized into one of four conditions: 1) Active cooking classes followed by meal kits and recipes, 2) Active cooking classes followed by no further instruction, 3) No cooking classes followed by meal kits and recipes, or 4) No intervention. Assessments will be conducted at baseline and following each phase.

DETAILED DESCRIPTION:
The proposed pilot study is a randomized trial to evaluate whether cooking classes produce greater gains in cooking skills, food agency, and cooking frequency than meal kits or no intervention. There will be three phases to the study intervention and four study conditions (as outlined below).

Phase 1- Cooking classes. All participants will attend 1 kitchen intensive session followed by 1 cooking class per week for 6 weeks

Phase 2- Meal Kits. Assigned participants will receive meal kit deliveries once per week for 6 weeks.

Phase 3- Recipes. Assigned participants will receive 5 healthy recipes by email once per week for 6 weeks. This phase was planned, but was canceled due to disruptions caused by the COVID-19 outbreak.

The investigators will randomize 64 students to one of four intervention conditions.

Group A (n=16) - Active cooking classes followed by meal kits and recipes Group B (n=16) - Active cooking classes followed by no further instruction Group C (n=16) - No cooking classes followed by meal kits and recipes Group D (n=16) - No intervention

Assessments will be conducted at baseline, and following each phase.

Cooking Classes: Subjects in the cooking class conditions will begin with a brief lecture on the day's lesson followed by a demonstration from the chef instructor. Subjects will then work with a partner to prepare the recipe with guidance from the chef instructor. All participants will receive printed copies of the weekly recipe(s). At the end of the class period all subjects will take part in a sensory experience led by the chef instructor in which they will observe the appearance, smell, taste, and texture, of the meal they have just prepared.

Meal Kits: With the meal delivery service, participants will get all the ingredients they need to make a meal as well as a recipe for the meal which includes step-by-step photos. They are then responsible for doing the actual cooking of the meal. Students will all receive kits for 3 meals per week from the same delivery service and will have the option to select meals that fit their dietary needs (vegetarian, gluten free, etc.). Meal kits are designed to serve two individuals therefore students should have enough food for six meals, though they will only need to cook three times. The service used is open to the public, therefore students who enjoyed the meal kit service could opt to continue service and pay for it themselves. However, students will be instructed to wait until study completion to do so.

Recipes: Recipes will be designed by the research team, which includes three registered dietitians and a trained chef. Students will receive recipes for five healthy meals per week. Participants will need to shop, budget, and plan on their own. Recipes will accommodate major dietary preferences including vegetarian and gluten-free.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at the University of Vermont living off campus independently (may have roommates but not live with a guardian)
* Ages 18-25
* Cooks dinner at home no more than 3x/week
* Access to a kitchen at home
* Availability during scheduled cooking classes/demonstrations

Exclusion Criteria:

* Students will be excluded from the study if they do not complete baseline data collection measures prior to the first class meeting.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lizzy F Pope, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Cooking +Meal Kits and Recipes: Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal.
  Following 6 weeks of cooking classes, participants will receive 6 weeks of home-delivered meal kits. Following 6 weeks of meal kits, participants will received 6 weeks of recipes. Both the meal kits and recipes will accommodate major dietary needs (vegan, gluten-free, etc.)
  Active Cooking + Meal Kits + Recipes: 6 cooking classes will be held every week for 6 consecutive weeks. The lessons are patterned after Dr. Amy Trubek's cooking pedagogy and will be tailored for those cooking for themselves for the first time. Classes begin with a brief lecture on the day's topic. Students will work in teams of 2 in the foods lab to actively practice skills and cook a meal. Students receive recipes and information sheets that cover pantry supplies, grocery lists, knife skills and cooking equipment. All students attend a 2 hour kitchen intensive demonstration as an orientation. After 6 weeks students receive 6 weeks of meal kits followed by 6 weeks of recipes.
- Active Cooking Only: Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal. Unlike the previous arm, no further instruction will be given once cooking classes end.
  Active cooking: Students receive the same cooking intervention and kitchen intensive orientation as described in the Active cooking + meal kits + recipes. However, once the 6 weeks of the cooking class have ended, there is no further intervention.
- Meal Kits and Recipes Only: Participants will receive weekly meal kit deliveries for 6 weeks.
Period: Overall Study
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits and Recipes Only | Control
Started | 18 | 16 | 9 | 10
Completed | 18 | 16 | 9 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control | Total
Number analyzed (Participants) | 18 | 16 | 9 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (1.33) | 20.9 (1.23) | 20.6 (.5) | 20.6 (.84) | 20.7 (1.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 13 | 7 | 9 | 41
  Male | 4 | 3 | 2 | 1 | 10
  Non-binary/ third gender | 1 | 0 | 0 | 0 | 1
  Prefer not to answer | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 14 | 14 | 9 | 10 | 47
  East Asian or Asian American | 2 | 0 | 0 | 0 | 2
  Latino or Hispanic American | 1 | 0 | 0 | 0 | 1
  Black, Afro-Caribbean, or African American | 0 | 1 | 0 | 0 | 1
  South Asian or Indian American | 1 | 0 | 0 | 0 | 1
  Bi-racial | 0 | 1 | 0 | 0 | 1
Relationship Status [Count of Participants; unit: Participants]
  Single | 18 | 14 | 8 | 10 | 50
  Living with partner | 0 | 2 | 1 | 0 | 3
Employment Status [Count of Participants; unit: Participants]
  10 - 20 hours per week | 5 | 3 | 4 | 2 | 14
  < 10 hours per week | 7 | 5 | 4 | 7 | 23
  No Employed | 6 | 8 | 1 | 1 | 16
University Standing [Count of Participants; unit: Participants]
  Junior | 8 | 4 | 2 | 4 | 18
  Senior | 7 | 12 | 7 | 6 | 32
  Other | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Diet Quality at Baseline and Change From Baseline
Description: Difference in diet quality change between groups from baseline, end of phase 1, and end of phase 2. Measured by Healthy Eating Index scores.
  The HEI includes 13 components that capture recommendations of the 2015-2020 Dietary Guidelines for Americans. There are two groupings of components:
  1. Adequacy components are encouraged. Higher scores reflect higher intakes.
  2. Moderation components should be limited. Higher scores reflect lower intakes. A higher total HEI score reflects higher diet quality as defined by the Dietary Guidelines for Americans.
  Components are weighted equally and assigned a score of either 5 or 10. Scores as summed to determine total score. Score range is 0 - 100.
  Adequacy Components:
  Total Fruits 5 Whole Fruits 5 Total vegetables 5 Greens and beans 5 Whole grains 10 Dairy 10 Total protein foods 5 Seafood and plant proteins 5 Fatty acids 10
  Moderation Components:
  Refined grains 10 Sodium 10 Added sugars 10 Saturated fats 10
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Cooking +Meal Kits and Recipes: Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal.
  Following 6 weeks of cooking classes, participants will receive 6 weeks of home-delivered meal kits.
- Meal Kits Only: Participants will receive weekly meal kit deliveries for 6 weeks.
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
score on a scale
  Baseline Score | 65.11 (3.17) | 61.84 (3.37) | 61.08 (4.49) | 67.84 (4.49)
  Phase 1 Score Change | -7.45 (3.09) | -3.52 (3.8) | -7.26 (4.37) | -4.71 (4.57)
  Phase 2 Score Change | -4.65 (3.37) | -2.07 (4.42) | -5.7 (4.55) | -4.56 (4.63)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = 0.91, Mixed Models Analysis

2. Secondary Outcome: Cooking and Food Practices at Baseline and Change From Baseline
Description: Cooking and Food Practices score at baseline and change at phase 1 and phase 2, will be measured by The Cooking and Food Provisioning Action Scale (CAFPAS) measures food preparation skills and capacities. The CAFPAS contains 28 items administered with a 7-point bipolar Likert scale. There are three subscales: Self-Efficacy (measures whether an individual thinks their cooking ability and skills are adequate), Attitude (measures an individual's affective stance towards food, cooking and provisioning in different areas), and Structure (measures the ways in which external factors can either hinder or support an individual's cooking and provisioning actions). Subscales are scored by coding responses from 1-7, reversing them as necessary, summing the items and dividing by the standard deviation of the sample population's scores on the subscale. The total CAFPAS score is the sum of the three subscales. The total score range is 3-196. A higher score is associated with improvement.
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Cooking Only: Participants will attend a weekly 2-hour cooking class to learn how to prepare meals. Participants cook and sample the meal at the end of class and the chef will walk them through a sensory exercise. At the end of each class, participants will be provided with the recipe for the next class and asked to create a timeline for the various steps of preparation. Participants will bring this timeline to class and discuss as a group before preparing the meal. Unlike the previous arm, no further instruction will be given once cooking classes end.
  .
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
score on a scale
  Baseline Score | 11.7 (.47) | 11.85 (.5) | 11.64 (.67) | 12.66 (.63)
  Phase 1 Score Change | 2.03 (.37) | 2.03 (.46) | .007 (.54) | .87 (.51)
  Phase 2 Score Change | -.40 (.38) | -.21 (.59) | 1.6 (.55) | .68 (.52)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = 0.03, Mixed Models Analysis

3. Secondary Outcome: Stress Level at Baseline and Change From Baseline
Description: The Perceived Stress Scale is a reliable and valid measure of perceived stress in adults including college students. Ten questions assess how often one perceives various forms of stress such as feeling unable to control important events, being upset by something unexpected, and feeling nervous. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
score on a scale
  Baseline Score | 19.28 (1.55) | 18.94 (1.65) | 20.33 (2.2) | 19.5 (2.09)
  Phase 1 Score Change | -2.56 (1.22) | 1.51 (1.52) | 1.0 (1.72) | 0.48 (1.71)
  Phase 2 Score Change | 2.64 (1.27) | -3.68 (1.96) | -4.20 (1.8) | -4.78 (1.72)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = 0.91, Mixed Models Analysis

4. Secondary Outcome: Breakfast Cooking Frequency at Baseline and Change From Baseline
Description: Breakfast cooking frequency was assessed at baseline and following each 6 week study phase using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: meals cooked
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
meals cooked
  Baseline | 1.78 (.43) | 1.75 (.46) | 2.67 (.61) | 4.4 (.58)
  Phase 1 Change | .78 (.50) | .31 (.61) | 0.44 (7.1) | -.31 (.70)
  Phase 2 Change | 1.42 (.52) | -.07 (7.9) | .12 (.74) | .33 (.71)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = .19, Mixed Models Analysis

5. Secondary Outcome: Lunch Cooking Frequency at Baseline and Change From Baseline
Description: Lunch cooking frequency was assessed at baseline and following each 6 week study phase using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: meals cooked
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
meals cooked
  Baseline | 1.33 (.40) | .75 (.42) | 2.44 (.56) | 2.9 (.53)
  Phase 1 Change | .33 (.39) | .90 (.48) | -.22 (.55) | .56 (.54)
  Phase 2 Change | .78 (.45) | .88 (.62) | .96 (.57) | .44 (.55)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = .77, Mixed Models Analysis

6. Secondary Outcome: Dinner Cooking Frequency at Baseline and Change From Baseline
Description: Dinner cooking frequency was assessed at baseline and following each 6 week study phase using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: Baseline, end of phase 1, and end of phase 2, up to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: meals cooked
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
Number analyzed (Participants) | 18 | 16 | 9 | 10
meals cooked
  Baseline | 2.7 (.40) | 3.38 (.42) | 4.11 (.56) | 4.7 (.53)
  Phase 1 Change | .78 (.45) | .23 (.54) | .11 (.63) | .84 (.62)
  Phase 2 Change | 1.45 (.47) | -.46 (.71) | .11 (.66) | .11 (.63)
Statistical Analysis 1: Comparison: Active Cooking +Meal Kits and Recipes vs Active Cooking Only vs Meal Kits Only vs Control; Test type: Superiority; p = .06, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline through phase 2 completion, an average of 12 weeks.
Arm/Group | Active Cooking +Meal Kits and Recipes | Active Cooking Only | Meal Kits Only | Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
The final planned 6-week intervention phase, Recipe Provision, was cancelled due to disruptions related to the COVID-19 pandemic. Following spring break, the university transitioned to remote instruction and the majority of the study participants moved back home to live with parents or guardians. As the study was designed to measure cooking behaviors and outcomes in a population of students preparing food independently, the study intervention and data collection could not continue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT04084028/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT04084028/ICF_001.pdf